CLINICAL TRIAL: NCT00948077
Title: A Single-Center, Open-Label, Randomized, Crossover Design Study to Evaluate the Effect of Dietary Status on Pharmacokinetic Profile of Orally Administered First-Line Anti-TB Drugs in Subjects With Pulmonary Tuberculosis
Brief Title: Pharmacokinetic Study for Anti-tuberculosis Drugs
Acronym: TBPK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Ming-Chih Yu, M.D./Chief, Taipei Medical University WanFang Hospital - Division of Pulmonary Medicine
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2009WFCRC-08; 98040
Record Dates: First submitted 2009-06-16; First posted 2009-07-29 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Pulmonary Tuberculosis
Keywords: tuberculosis; pharmacokinetic; first-line drugs
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — isoniazid, pyrazinamide, rifampin drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Active Comparator): Study agents (Rifater+EMB) will be given approximately 45 minutes "prior to the breakfast."
  Interventions: Drug: Rifater and EMB
- Treatment B (Experimental): Study agents (Rifater+EMB) will be given approximately 45 minutes "after the breakfast is finished."
  Interventions: Drug: Rifater and EMB

INTERVENTIONS:
Drug: Rifater and EMB — The main difference between Treatment A and Treatment B is the time of taking drugs, so the intervention of this study belongs to a behavioral intervention.
  The patients assigned randomly the Arm "Treatment A" on the fifth day will be switched to the Arm "Treatment B" on the sixth day. On the other hand, the patients assigned randomly the Arm "Treatment B" on the fifth day will be switched to the Arm "Treatment A" on the sixth day. The flow of intervention is drawn as below.
  Treatment A (5th day) ---> Treatment B (6th day) ; Treatment B (5th day) ---> Treatment A (6th day)

SUMMARY:
The purpose of this study is to evaluate the effect of food on pharmacokinetic profile of multiple doses orally administered first-line anti-tuberculosis drugs in subjects with pulmonary tuberculosis.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, two way crossover design, pharmacokinetics study.

1. Treatment A: study agents (Rifater+EMB) will be given approximately 45 minutes prior to breakfast.
2. Treatment B: study agents (Rifater+EMB) will be given approximately 45 minutes after the breakfast is finished.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 20 years
2. Karnofsky score of > 50
3. Clinical and radiographic signs and symptoms consistent with pulmonary TB determined by the investigator.
4. A documented positive microbiology diagnosis results which indicate highly suspected pulmonary tuberculosis.
5. Anti-TB drugs treatment with of ethambutol, isoniazid, rifampin and pyrazinamide.
6. Willing to be hospitalized per standard of care for at least 6 days from first does of anti-TB drugs administered.
7. Start anti-TB chemotherapy for at least 2 days prior to participate in the study.
8. The subject is able to understand and comply with protocol requirements, and follow the instructions and protocol-stated restrictions.
9. Only subjects who have provided signed and dated written informed consent will be included.

Exclusion Criteria:

1. Previously treated for MDR-TB, XDR-TB or likely to require surgical procedure for management of TB
2. Alcohol or drug abuse that would interfere with the ability to meet study requirements (in the opinion of investigator)
3. Concomitant disorders or conditions for which ethambutol, isoniazid, rifampin or pyrazinamide are contraindicated.
4. Unable to meet selected safety criteria obtained at screening (Laboratory parameters, etc.)
5. Women who are Pregnant or breastfeeding during the study period.
6. Subjects with a known allergy to study drugs
7. In the opinion of the investigator to be unsuitable for study participation for any reason.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The maximum concentration (Cmax)of first-line TB drugs | Before and 1, 2, 4, 6 and 10 hours after dosing

SECONDARY OUTCOMES:
N-acetyltransferase 1 and 2 (NAT 1 and 2), which effects the metabolism of anti-TB drugs, would be examined. | Before taking the anti-TB drugs on the fifth day

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih MC Yu, M.D., Principal Investigator — Taipei Medical University- Wan Fang Hospital
Locations (1):
- Taipei Medical University- Wan Fang Hospital, Taipei, Taiwan